CLINICAL TRIAL: NCT03159442
Title: A Phase I, Single Centre, Randomised, Single Blind, Placebo-Controlled Study to Investigate the Safety, Tolerability and Pharmacokinetics of Multiple Ascending Doses of Inhaled AZD8871 in Healthy Male Japanese Subjects.
Brief Title: Safety, Tolerability and Pharmacokinetics of Multiple Ascending Doses of AZD8871 in Healthy Male Japanese Subjects
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: AstraZeneca (Industry)
Collaborators: Parexel (Industry); Industrias Farmacéuticas Almirall S.A. (Unknown); The Doctors Laboratory Ltd (Industry); Covance (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: D6640C00005; 2017-000890-35 (EudraCT Number)
Record Dates: First submitted 2017-05-17; First posted 2017-05-18 (Actual); Last update posted 2017-10-25 (Actual); Status verified 2017-10

CONDITIONS: Chronic Obstructive Pulmonary Disease - COPD
Keywords: Chronic obstructive pulmonary disease (COPD); Asthma; AZD8871; muscarinic receptor antagonist and β2 adrenoceptor agonist (MABA); Phase I; Safety; Tolerability; Pharmacokinetics; long-acting muscarinic antagonist (LAMA); long-acting β2-agonist (LABA); Japanese
MeSH Terms: conditions — Pulmonary Disease, Chronic Obstructive; Asthma | interventions — AZD-8871

STUDY DESIGN:
Intervention Model Description: Single center, randomized, single blind, placebo-controlled study.
Who Masked: Participant
Masking Description: This study is single-blind with regards to treatment (AZD8871 or placebo) at each dose level. However, the study centre staff are also blinded only during the clinical conduct of a given cohort prior to the respective safety review committee meeting (SRC).
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (3):
- Cohort 1 (Experimental): Multiple inhaled doses of AZD8871 will be administered via single dose DPI. Each subject will receive 300 μg AZD8871 or placebo. This dose will be given as 1 inhalation from the 300 μg AZD8871 or placebo inhaler.
  Single inhaled dose of AZD8871 or placebo will be administered on Day 1 and then single once daily inhalations of AZD8871 or placebo will be administered for 12 days from Day 5 until Day 16.
  Interventions: Drug: AZD8871; Drug: Placebo
- Cohort 2 (Experimental): Multiple inhaled doses of AZD8871 will be administered via single dose DPI. Each subject will receive 600 μg AZD8871 as 1 inhalation from the 600 μg AZD8871 or placebo inhaler.
  Single inhaled dose of AZD8871 or placebo will be administered on Day 1 and then single once daily inhalations of AZD8871 or placebo will be administered for 12 days from Day 5 until Day 16.
  Dose escalation to 600 μg dose will be done only after the SRC has determined the adequacy of the dose to be given.
  Interventions: Drug: AZD8871; Drug: Placebo
- Cohort 3 (Experimental): Multiple inhaled doses of AZD8871 will be administered via single dose DPI. Each subject will receive 900 μg AZD8871 as 1 inhalation from the 300 μg AZD8871 inhaler and 1 inhalation from the 600 μg AZD8871 inhaler, or placebo as 2 inhalations from 2 different placebo inhalers.
  Single inhaled dose of AZD8871 or placebo on Day 1 and then single once daily inhalations of AZD8871 or placebo will be administered for 12 days from Day 5 until Day 16.
  Dose escalation to the 900 μg dose will be done only after the SRC has determined the adequacy of the dose to be given.
  Interventions: Drug: AZD8871; Drug: Placebo

INTERVENTIONS:
Drug: AZD8871 — Powder for inhalation administered via single dose DPI 300 and 600 µg/inhalation.
Drug: Placebo — Powder for inhalation administered via single dose DPI

SUMMARY:
AZD8871 is a new chemical entity possessing long-acting dual-pharmacology (muscarinic receptor antagonist and β2 adrenoceptor agonist [MABA]) in a single molecule. This type of agent presents a novel approach to the treatment of chronic obstructive pulmonary disease (COPD) and potentially asthma (in combination with an inhaled corticosteroid). AZD8871 is being developed for inhalation, formulated with alpha lactose monohydrate and delivered by dry powder inhaler (DPI) that allows delivery of a single dose of the study drug.

The primary objective is to investigate the safety and tolerability of AZD8871 at steady state in healthy male Japanese subjects.

DETAILED DESCRIPTION:
This is a Phase I, single centre, randomised, single blind, placebo-controlled study to investigate the safety, tolerability and pharmacokinetics (PK) of single and multiple ascending doses of inhaled AZD8871 in healthy male Japanese subjects.

All subjects will sign an Informed Consent Form before starting any study-related procedures.

Twenty-four healthy subjects, aged 20 to 55 years, will participate in 3 cohorts. All subjects will be admitted to the unit the day preceding the 1st dose and will be housed in the unit until 96 hours (4 days) post last dose of investigational medicinal product (IMP) (Day 20).

Eight subjects will participate in each cohort and will receive either AZD8871 or placebo, randomised 3:1 (6 subjects to receive AZD8871:2 subjects to receive placebo). Each subject will only be dosed in 1 cohort. The study design allows a gradual escalation of dose (Cohorts 2 and 3) with intensive safety monitoring to ensure the safety of the subjects.

In Cohort 1, subjects will receive only a single dose of AZD8871 300 µg or placebo on Day 1, followed by once daily dosing on Days 5 to 16. The dosing schedule of all cohorts will be single dose of IMP (active or placebo) on Day 1, followed by once daily dosing on Days 5 to 16. Within 5 to 7 days of discharge from the unit, there will be two follow-up visits.

Following each cohort, a maximum dose of 2 times the dose administered in the previous cohort will be considered for the subsequent cohort. However, the planned dose for Cohort 2 is 600 µg and for Cohort 3 is 900 µg. Dosing of Cohorts 2 and 3 will be preceded by a SRC meeting, which will confirm the adequacy of the planned doses. A minimum of 5 subjects on active treatment need to complete dosing per cohort in order to proceed to the next dose level.

The total duration of the study for each subject will be approximately 58 days (from Screening [up to -28 days before randomization] to Final Follow up visit [Day 30]).

ELIGIBILITY:
Inclusion Criteria:

1. Provision of written informed consent prior to any study related procedures, including withdrawal of medications.
2. Male Japanese subjects aged 20 to 55 years, inclusive at Screening.
3. Body mass index (BMI) calculated as weight in kg/height in m2 from >= 18 to <= 30 kg/m2 and weight >= 50 kg at Screening.
4. Healthy, free from any clinically significant disease/conditions (including all cardiovascular conditions), as determined by medical history, physical examination, clinical laboratory testing, 12-lead ECG findings at Screening and admission to the unit.
5. Spirometry readings (Forced Expiratory Volume in 1 second and Forced Vital Capacity) to be >= 80% of predicted value calculated using equations at Screening (Quanjer et. al. 2012).
6. Normal blood pressure (BP) (defined as systolic BP >= 90 and <= 140 mmHg and diastolic BP >= 50 and <= 90 mmHg) at Screening and admission to the unit, measured after resting in supine position for at least 10 minutes.
7. Normal heart rate (HR) (defined as HR >= 45 and <= 90) measured after resting in supine position for at least 10 minutes at Screening and admission to the unit.
8. Negative hepatitis B surface antigen (HBsAg), hepatitis B core (HBc) antibody (IgM), hepatitis C antibody and human immunodeficiency virus (HIV) I and II antibodies at Screening.
9. Negative drugs of abuse and alcohol tests at Screening and at admission to the unit.
10. Willing and able to comply with study specific procedures and restrictions.

Exclusion Criteria:

1. Involvement in the planning and/or conduct of the study (applies to both AstraZeneca staff and/or staff at the study site)
2. Surgical history clinically relevant for the purpose of the study or any clinically significant illness, medical/surgical procedure or trauma within 4 weeks of Screening.
3. History of malignancy of any organ system, treated or untreated within the past 5 years, with the exception of localised basal cell carcinoma of the skin.
4. Current smokers, or a smoking history during the last 6 months or total smoking history of more than 10 pack years. Use of electronic cigarettes or other forms of nicotine, current use or use within the last 6 months.

   Note: Pack years are calculated by dividing the number of cigarettes smoked per day by 20 (the number of cigarettes per pack) and multiplying tis figure by the number of years a person has been smoking. For example, a person who smoked 40 cigarettes a day and has been smoking for 10 years would have a 20 pack-year smoking history (40 cigarettes per day at 20 cigarettes per pack =2; 2 x 10 years of smoking =20 pack-year history).
5. Prolonged QTcF corrected using Fredericia's formulae) interval, > 450 ms at Screening, or family history of long QT syndrome.
6. Any clinically significant abnormalities in rhythm, conduction or morphology noted on physical examination, ECG or telemetry recording, prior to randomisation.
7. History of excessive use or abuse of alcohol within the past 2 years, defined as: subjects consuming more than 21 (male subjects) units of alcohol a week (1 unit = 1 glass of wine (125 mL) = 1 measure of spirits = half pint of beer).
8. History of drug abuse within the past 2 years prior to Screening.
9. Donation or loss of > 400 ml blood and plasma within the previous 3 months prior to Screening.
10. History or presence of severe allergy/hypersensitivity or ongoing allergy/hypersensitivity to any drug, as judged by the Investigator or history of hypersensitivity to drugs pharmacologically related to study drug.
11. PR (PQ) interval shortening < 120 ms (PR > 110 ms but < 120 ms is acceptable if there is no evidence of ventricular pre-excitation) at Screening.
12. PR (PQ) interval prolongation (> 240 ms), intermittent second (Wenckebach block while asleep is not exclusive), or third degree AV block, or AV dissociation at Screening.
13. Persistent or intermittent complete bundle branch block, incomplete bundle branch block.
14. Intraventricular conduction delay with QRS (onset of ventricular depolarization) > 110 ms at Screening.

    Note: Subjects with QRS > 110 ms but < 115 ms are acceptable if there is no evidence of ventricular hypertrophy or pre-excitation.
15. Subject who does not agree to follow instructions to avoid partner pregnancy.
16. Subject who is not able to adhere to the restrictions on prior and concomitant medications.
17. Administered any investigational drug within 3 months prior to first dosing in this study or within the equivalent time of 5 half lives of receiving the last IMP administration, whichever is longer, or on an extended Follow up after receiving an IMP.
18. Subjects unable to communicate reliably with the Investigator, even with the help of an interpreter.
19. Vulnerable subjects, e.g., kept in detention, protected adults under guardianship, trusteeship, or committed to an institution by governmental or juridical order.
20. Subjects who failed any Screening procedures will not be included in the study.
21. Subjects with psychiatric disease with limitations to follow instructions in regards of study procedures.
22. Subjects with serum potassium values < 3.5 mmol/L at Screening and on repeat testing.

    Note: Potassium replacement and repeat testing is allowed if serum potassium concentration was < 3.5 mmol/L at Screening.
23. Any laboratory abnormality or suspicion of any clinically relevant disease or disorder (on history or examination), including uncontrolled diabetes, which, in the opinion of the Investigator, may either put the subject at risk because of participation in the study, or influence the results or the subject's ability to participate in the study, or any other safety concern in the opinion of the Investigator.

Ages: 20 Years to 55 Years | Sex: Male | Healthy Volunteers: Yes
Age Groups: Adult
Gender Based: Yes — Male Japanese subjects aged 20 to 55 years, inclusive at Screening.
  A Japanese subject is defined as a subject who was born in Japan and has 2 Japanese biological parents and 4 Japanese grandparents, as confirmed by interview. The subject should not have been living outside of Japan for more than 5 years at the time of the Screening visit. The subjects should not have had a significant change in lifestyle or diet since leaving Japan.
Enrollment: 25 (Actual)
Dates: Start 2017-06-19 (Actual); Primary Completion 2017-10-13 (Actual); Study Completion 2017-10-13 (Actual)

PRIMARY OUTCOMES:
Adverse events. | From time of ICF to Day 30 (end of follow-up period)
  Recording adverse events. An AE is the development of an undesirable medical condition or the deterioration of a preexisting medical condition following or during exposure to a pharmaceutical product, whether or not considered causally related to the product. An undesirable medical condition can be symptoms (e.g., nausea, chest pain), signs (e.g., tachycardia, enlarged liver) or the abnormal results of an investigation (e.g., laboratory findings, ECG). In clinical studies, an AE can include an undesirable medical condition occurring at any time, including run-in or washout periods, even if no study treatment has been administered.
Concomitant medication. | Change from screening up to follow-up period (Day 30 +/- 1)
  Recording concomitant medications. Any concomitant medication or therapy given to the subject during the study conduct will be recorded.
Physical examination. | Change from screening up to follow-up period (Day 30 +/- 1)
  A full physical examination will include the examination of the following: general appearance, eyes, ears, nose, throat, chest/respiratory, heart/cardiovascular, gastrointestinal/liver, musculoskeletal/extremities, dermatological/skin, thyroid/neck, lymph nodes, neurological/psychiatric.
  A brief physical examination will include assessment of the following: skin, lungs, cardiovascular system and abdomen (liver and spleen).
  A complete physical examination will be performed at the Screening and Follow-up visit.
  Only relevant findings detected will be recorded in the physical examination findings.
Vital signs. | Change from screening up to follow-up period (Day 30 +/- 1)
  Recording vital signs. Systolic and diastolic blood pressure (in mmHg) will be measured after at least 10 minutes (can be reduced to 5 minutes at collection time points within the 1st hour after dosing) resting, and also, before taking any blood sample and conducting any spirometry. Measurements will be carried out with subject in the supine position and preferably always on the same arm.
  Subject's oral body temperature will be measured at each vital signs collection.
Number of clinically relevant new findings or worsening of a pre-existing findings as assessed by Hematology. | Change from screening up to follow-up period (Day 30 +/- 1)
  Haematocrit, hemoglobin, erythrocytes (red blood cells), mean corpuscular volume (MCV), mean corpuscular haemoglobin (MCH), mean corpuscular haemoglobin concentration (MCHC), leucocytes (white blood cells), differential blood count (neutrophils, lymphocytes, monocytes, eosinophils and basophils) and thrombocytes (platelets)
Number of clinically relevant new findings or worsening of a pre-existing findings as assessed by Clinical chemistry. | Change from screening up to follow-up period (Day 30 +/- 1)
  Electrolytes: sodium, potassium, calcium, chloride and inorganic phosphorus. Enzymes: AST, ALT, ALP, GGT, LDH, creatine kinase. Substrates: glucose (fasting), total cholesterol, triglycerides, creatinine, TBL, total protein, albumin, uric acid, urea and BUN.
  Endocrinology: T4, TSH. Viral serology: HIV I and II antibodies, hepatitis C antibodies, HBsAg, HBc. Coagulation: INR, PT, aPTT.
ECG. | Change from screening up to follow-up period (Day 30 +/- 1)
  A 12-lead ECG will be obtained after the subject rested in the supine position for at least 10 minutes (can be reduced to 5 minutes at collection time points within the first hour after dosing; using the sites own ECG machines when not performing dECGs and using the same machine as the dECGs when time points coincide).
2-lead real-time telemetry ECG. | Change from screening up to follow-up period (Day 30 +/- 1)
  Recording telemetry findings. A 2-lead real-time telemetry ECG will be performed for at least 4 hours on Day 1 and then on Days 1, 10 and 16 from 30 minutes predose until 24 hours postdose.
Number of clinically relevant new findings or worsening of a pre-existing findings as assessed by urinalysis report. | Change from screening up to follow-up period (Day 30 +/- 1)
  pH, blood, leucocytes, protein, glucose, bilirubin, urine bilirubin, ketones and nitrites.
  If clinically relevant abnormalities are detected (positive result in dipstick), microscopy (RBC, WBC and cast [hyaline, granular and cellular]).

SECONDARY OUTCOMES:
Observed maximum concentration, taken directly from the individual concentration-time curve (Cmax) of AZD8871 and its metabolites. | Day 1 and Day 16
  Observed maximum concentration.
Time to reach maximum concentration, taken directly from the individual concentration-time curve (tmax) of AZD8871 and its metabolites. | Day 1 and Day 16
  Time to reach maximum concentration.
Terminal half-life (t½λz) of AZD8871 and its metabolites. | Day 1 and Day 16
  Terminal half-life, estimated as (ln2)/λz.
Area under the plasma concentration-curve from time zero to 24 hours post-dose (AUCτ) of AZD8871 and its metabolites. | Day 1 and Day 16
  Area under the plasma concentration-curve from time zero to 24 hours post-dose
Area under the concentration-time curve from time zero extrapolated to infinity (AUC) of AZD8871 and its metabolites. | Day 1
  Area under the concentration-time curve from time zero extrapolated to infinity. AUC is estimated by AUC0-last + C-last/λz where C-last is the last observed quantifiable concentration.
Apparent clearance for parent drug (CL/F) estimated as dose divided by AUC of AZD8871 and its metabolites. | Day 1 and Day 16
  Apparent clearance for parent drug estimated as dose divided by AUC.
Apparent volume of distribution for parent drug at terminal phase (Vz/F) of AZD8871 and its metabolites. | Day 1
  Apparent volume of distribution for parent drug at terminal phase (extravascular administration), estimated by dividing the apparent clearance (CL/F) by λz.
Accumulation ratio for Cmax (Rac (Cmax)) of AZD8871 and metabolites after repeated administration. | Day 16
  Accumulation ratio for Cmax estimated as Cmax on Day 16/Cmax on Day 1.
Accumulation ratio for AUCτ (RacAUCτ) of AZD8871 and metabolites after repeated administration. | Day 16
  Accumulation ratio for AUCτ estimated as AUCτ on Day 16/AUCτ on Day 1.

CONTACTS AND LOCATIONS:
Overall Officials: Muna Albayaty, MBChB, MSc, MFPM, Study Chair — Parexel
Locations (1):
- Research Site, London, United Kingdom

IPD SHARING:
Plan to Share IPD: Undecided

REFERENCES:
- [Derived] Balaguer V, Albayaty M, Jimenez E, Wahlby-Hamren U, Astbury C, Seoane B, Malice MP, Lei A, Aggarwal A, Psallidas I. Navafenterol (AZD8871) in healthy volunteers: safety, tolerability and pharmacokinetics of multiple ascending doses of this novel inhaled, long-acting, dual-pharmacology bronchodilator, in two phase I, randomised, single-blind, placebo-controlled studies. Respir Res. 2020 Sep 9;21(Suppl 1):212. doi: 10.1186/s12931-020-01474-1. PMID 32907575